CLINICAL TRIAL: NCT02703597
Title: Social Influence Strategies During a Web-based Smoking Prevention Intervention for Adolescents
Brief Title: Smoking Prevention Through Social Connections Among Adolescents - ASPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2015-0995; NCI-2016-00554 (Registry Identifier: NCI CTRP); 1K99DA044277-01A1 (NIH); IRB201903082 (Other: University of Florida IRB); R00DA044277 (NIH)
Record Dates: First submitted 2016-03-04; First posted 2016-03-09 (Estimated); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-09

CONDITIONS: Tobacco Use Behavior
Keywords: Tobacco; Curiosity; Tobacco Cessation; Tobacco Prevention; Health improvement; Smoking prevention interactive experience; ASPIRE; Games for health; Surveys; Questionnaires; Interviews; Focus Group
MeSH Terms: conditions — Exploratory Behavior; Tobacco Use Cessation | interventions — Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will not know if they are receiving the intervention to be tested or the comparative intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASPIRE Group (Experimental): Participants engage in up to five 70-minute sessions of ASPIRE spread over a period of 5 weeks. Each session completion has a window of 2 weeks, taking into account site availability, presence of students, holidays, and site resources. During ASPIRE use, participants face a screen and individually watch videos and engage in computer-based activities related to the negative effects of tobacco. At baseline, after 3 sessions, following the last session of the intervention, and about one month after the intervention has ended, participants complete psychosocial surveys and social network surveys. Baseline survey again completed. About one month after assessment 4, this group receives a 5th assessment followed by a hybrid version of the GSA-ASPIRE-Network program (moderated by Kahoot!). The group receives additional assessments after 3 sessions, following the last session of the program, and about one month after the program has ended (assessment 8).
  Interventions: Behavioral: Surveys; Behavioral: ASPIRE
- GSA-ASPIRE-Network Group (Experimental): Participants engage in five 70-minute sessions of ASPIRE conducted over a period of 5 weeks, with 2 booster sessions. Each session completion has a window of 2 weeks, taking into account site availability, presence of students, holidays, and site resources. ASPIRE use is coupled with game-based social activities (GSAs). ASPIRE use, participants watch videos and engage in activities on the same computer. Each session, participants will alternate between 10 minutes of ASPIRE use and 5-minute GSAs. Participants engage in the paper-based GSAs as a team and collaborate as they complete the activities. The GSAs contain games about the effects of tobacco. Groups are allocated based on adolescents' network of friendships. At baseline, after 3 sessions, following the last session of the intervention, and about one month after the intervention has ended (assessment 4), participants complete psychosocial surveys and social network surveys.
  Interventions: Behavioral: Surveys; Behavioral: GSA-ASPIRE-Network

INTERVENTIONS:
Behavioral: Surveys — Surveys include questions related to tobacco use behavior and attitude toward tobacco, as well as demographic and personality questions. Psychosocial surveys and social network surveys are also completed to capture adolescents' network of friends and opinion leaders.
  Other Names: Questionnaires
Behavioral: ASPIRE — Participants engage in four to five 70-minute sessions of ASPIRE spread over a period of 4 weeks. During ASPIRE use, participants face a screen and individually watch videos and engage in computer-based activities related to the negative effects of tobacco.
  Arms: ASPIRE Group
Behavioral: GSA-ASPIRE-Network — In groups, participants engage in four to five 70-minute sessions of ASPIRE conducted over a period of 4 weeks. However, during each session, ASPIRE use is coupled with game-based social activities (GSAs). During ASPIRE use, participants watch videos and engage in computer-based activities on the same computer screen. Also, in groups, participants engage in the paper-based GSAs as a team and collaborate as they complete the activities. The GSAs contain games about the effects of tobacco. Groups are allocated based on adolescents' network of friendships.
  Arms: GSA-ASPIRE-Network Group

SUMMARY:
The central hypothesis of this study is that the addition of social influence strategies to a web-based program called ASPIRE will boost its success in lowering intention to use tobacco among adolescents and experiencing stronger positive social influence. The study will involve a nested group randomized controlled trial with adolescents from after-school programs and schools (e.g., the PK Yonge school) in Florida.

ELIGIBILITY:
Inclusion Criteria:

* All participants must be of ages 11 through 18 (11 and 18 included; age group for adolescents adopted by several National Institutes of Health)
* Are members of after school program or school
* All participants will be English speaking
* Adolescents with developmental disability, mental or physical, are not excluded from the study. However, they will only be able to participate if (1) they understand the information presented to them in the consent document, and (2) they believe they are capable to engage in the board game, use the internet, and answer survey questions.
* Pregnant adolescents will be eligible to participate in the research study as requested by the NIH based on 2 principles that will be discussed at time of consent.

Exclusion Criteria:

-When participants don't meet the inclusion criteria

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 393 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-03-16 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Georges Khalil, MPH, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khalil G, Ramirez E, Khan M, Zhao B, Ribeiro N, Balian P. Risk Perception and Knowledge Following a Social Game-Based Tobacco Prevention Program for Adolescents: Pilot Randomized Comparative Trial. JMIR Serious Games. 2024 Nov 5;12:e63296. doi: 10.2196/63296. PMID 39499912

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: after school programs
Groups:
- ASPIRE Group: Participants engage in up to five 70-minute sessions of ASPIRE spread over a period of 5 weeks. Each session completion has a window of 2 weeks, taking into account site availability, presence of students, holidays, and site resources. During ASPIRE use, participants face a screen and individually watch videos and engage in computer-based activities related to the negative effects of tobacco. At baseline, after 3 sessions, following the last session of the intervention, and about one month after the intervention has ended, participants complete psychosocial surveys and social network surveys. Baseline survey again completed. About one month after assessment 4, this group receives a 5th assessment followed by a hybrid version of the GSA-ASPIRE-Network program (moderated by Kahoot!). The group receives additional assessments after 3 sessions, following the last session of the program, and about one month after the program has ended.
  Surveys: Surveys include questions related to tobacco use behavior and attitude toward tobacco, as well as demographic and personality questions. Psychosocial surveys and social network surveys are also completed to capture adolescents' network of friends and opinion leaders.
  ASPIRE: Participants engage in four to five 70-minute sessions of ASPIRE spread over a period of 4 weeks. During ASPIRE use, participants face a screen and individually watch videos and engage in computer-based activities related to the negative effects of tobacco.
- GSA-ASPIRE-Network Group: Participants engage in five 70-minute sessions of ASPIRE conducted over a period of 5 weeks, with 2 booster sessions. Each session completion has a window of 2 weeks, taking into account site availability, presence of students, holidays, and site resources. ASPIRE use is coupled with game-based social activities (GSAs). ASPIRE use, participants watch videos and engage in activities on the same computer. Each session, participants will alternate between 10 minutes of ASPIRE use and 5-minute GSAs. Participants engage in the paper-based GSAs as a team and collaborate as they complete the activities. The GSAs contain games about the effects of tobacco. Groups are allocated based on adolescents' network of friendships. At baseline, after 3 sessions, following the last session intervention, and about one month after intervention, participants complete psychosocial surveys and social network surveys.
  Surveys: Surveys include questions on tobacco use behavior, attitude toward tobacco, and demographic and personality questions. Psychosocial surveys and social network surveys are also completed to capture adolescents' network of friends and opinion leaders.
  GSA-ASPIRE-Network Group: Participants engage in 4-5 weekly 70-minute ASPIRE sessions over 4 weeks, coupled with game-based social activities (GSAs). In groups, they watch videos, do computer activities, and collaborate on paper-based GSAs, which focus on tobacco's effects. Groups are formed based on adolescents' friendships.
Period: Assignment to Baseline
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 153; 7 after school programs | 240; 8 after school programs
Completed | 136; 7 after school programs | 224; 8 after school programs
Not Completed | 17; 0 after school programs | 16; 0 after school programs
Not completed — Lost to Follow-up | 17 | 16
Period: Baseline to First Post-test
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 136; 7 after school programs | 224; 8 after school programs
Completed | 75; 7 after school programs | 132; 8 after school programs
Not Completed | 61; 0 after school programs | 92; 0 after school programs
Not completed — Lost to Follow-up | 61 | 92
Period: First Post-test to First Follow-up
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 75; 7 after school programs | 132; 8 after school programs
Completed | 70; 7 after school programs | 71; 7 after school programs
Not Completed | 5; 0 after school programs | 61; 1 after school programs
Not completed — Lost to Follow-up | 5 | 3
Not completed — Site drop out | 0 | 58
Period: Recruitment Period for Assessment 5
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 70; 7 after school programs | 71; 7 after school programs
Completed | 54; 4 after school programs (4 sites agreed to participate in this stage of the trial.) | 0; 0 after school programs
Not Completed | 16; 3 after school programs | 71; 7 after school programs
Not completed — Withdrawal by Site | 16 | 0
Not completed — Were not expected to participate in this stage as per protocol | 0 | 71
Period: Recruitment to Assessment 5
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 54; 4 after school programs | 0; 0 after school programs (This group was not expected to participate in data collection at this point, as per the protocol.)
Completed | 54; 4 after school programs | 0; 0 after school programs (This group was not expected to participate in data collection at this point, as per the protocol.)
Not Completed | 0; 0 after school programs | 0; 0 after school programs
Period: Assessment 5 to Second Post-test
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Started | 54; 4 after school programs | 0; 0 after school programs (This group was not expected to participate in data collection at this point, as per the protocol.)
Completed | 27; 4 after school programs | 0; 0 after school programs (This group was not expected to participate in data collection at this point, as per the protocol.)
Not Completed | 27; 0 after school programs | 0; 0 after school programs
Not completed — Lost to Follow-up | 27 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group | Total
Number analyzed (Participants) | 153 | 240 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.09 (1.50) | 13.36 (1.36) | 13.26 (1.42)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed differs from overall because 74 participants did not answer the question.
  Participants
    number analyzed (Participants) | 133 | 186 | 319
    Female | 70 | 93 | 163
    Male | 63 | 93 | 156
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19 | 42 | 61
  Not Hispanic or Latino | 117 | 151 | 268
  Unknown or Not Reported | 17 | 47 | 64
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 5 | 6
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 103 | 109 | 212
  White | 8 | 52 | 60
  More than one race | 19 | 19 | 38
  Unknown or Not Reported | 19 | 47 | 66
Susceptible to using tobacco [Count of Participants; unit: Participants] — Using the original measure of susceptibility while considering several tobacco products including e-cigarettes, cigarettes, cigars, hookah, and chewing tobacco. Pierce JP, Choi WS, Gilpin EA, Farkas AJ, Merritt RK. Validation of susceptibility as a predictor of which adolescents take up smoking in the United States. Health psychology. 1996 Sep;15(5):355. Population: The row population differs from the overall number because some participants did not answer these survey questions.
  Participants
    number analyzed (Participants) | 136 | 229 | 365
    (all) | 80 | 132 | 212

OUTCOME MEASURES:

1. Primary Outcome: Susceptibility to Vaping
Description: During the course of the study surveys reviewed. This outcome was measured using a binary form of the susceptibility to vaping scale, which aims at measuring intention to vape. Scores were 0 (non-susceptible) or 1 (susceptible). A score of 1 has a worse value than a score of 0.
Time Frame: 4 weeks; Note that each survey completion has a window of 2 weeks, taking into account site availability, presence of students, holidays, and site resources.
Population: All collected data for this pre-specified Primary Outcome Measure is summarized and reported in this table. The number of participants analyzed differs from overall because not all participants answered the outcome measure survey questions.
Measure: Count of Participants; unit: Participants
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Number analyzed (Participants) | 137 | 229
Participants | 66 | 118
Statistical Analysis 1: Comparison: ASPIRE Group vs GSA-ASPIRE-Network Group; Hypothesis: Participants in the GSA-ASPIRE-Network Group will be more likely to decrease in susceptibility to vaping than participants in the ASPIRE group. The statistical analysis was conducted for 10 out of the 15 participating sites, to avoid bias with respect to the sites that participated in different conditions (i.e., 1 site in a school classroom during class time and 4 sites in the summer camp during summer time); Test type: Superiority; p = 0.80, Mixed Models Analysis; Odds Ratio (OR) = 1.15, 95% CI 2-sided [0.32 to 4.20]
Statistical Analysis 2: Comparison: ASPIRE Group vs GSA-ASPIRE-Network Group; Hypothesis: Participants in both arms will decrease in susceptibility to vaping over time. The statistical analysis was conducted for 10 out of the 15 participating sites, to avoid bias with respect to the sites that participated in different conditions (i.e., 1 site in a school classroom during class time and 4 sites in the summer camp during summer time); Test type: Superiority; p < 0.01, Mixed Models Analysis; Odds Ratio (OR) = 0.17, 95% CI 2-sided [0.06 to 0.43]

2. Primary Outcome: Susceptibility to Using Conventional Tobacco
Description: During the course of the study surveys reviewed. This outcome was measured using a binary form of the susceptibility to smoking scale, which aims at measuring intention to use conventional tobacco. Scores were 0 (non-susceptible) or 1 (susceptible). A score of 1 has a worse value than a score of 0. The measure combines susceptibility to using cigarettes, cigars, hookah, and chewing tobacco.
Time Frame: as for outcome 1
Population: All collected data for this pre-specified Primary Outcome Measure is summarized and reported in this table. The number of participants analyzed differs from overall because not all participants answered the outcomes measure survey questions.
Measure: Count of Participants; unit: Participants
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
Number analyzed (Participants) | 136 | 229
Participants | 63 | 106
Statistical Analysis 1: Comparison: ASPIRE Group vs GSA-ASPIRE-Network Group; Hypothesis: Adolescents who participated in the GSA-ASPIRE-Network group will be more likely to decrease in susceptibility to using conventional tobacco than adolescents who participated in the ASPIRE group. The statistical analysis was conducted for 10 out of the 15 participating sites, to avoid bias with respect to the sites that participated in different conditions (i.e., 1 site in a school classroom during class time and 4 sites in the summer camp during summer time); Test type: Superiority; p = 0.70, Mixed Models Analysis; Odds Ratio (OR) = 0.76, 95% CI 2-sided [0.16 to 3.49]
Statistical Analysis 2: Comparison: ASPIRE Group vs GSA-ASPIRE-Network Group; Hypothesis: Participants in both arms will decrease in susceptibility of using conventional tobacco over time. The statistical analysis was conducted for 10 out of the 15 participating sites, to avoid bias with respect to the sites that participated in different conditions (i.e., 1 site in a school classroom during class time and 4 sites in the summer camp during summer time); Test type: Superiority; p < 0.01, Mixed Models Analysis; Odds Ratio (OR) = 0.13, 95% CI 2-sided [0.04 to 0.40]

ADVERSE EVENTS:
Time Frame: 4 months
Description: At each session of data collection or intervention, the study staff were asked to record any adverse event that may occur, including a brief explanation of the event, when it occurred, the date of the event, description of what occurred, actions taken by research staff, planned follow up (if any), the intervention group/study arm of the affected participant, whether the event appears to be related to the intervention, and whether the participant will continue in the study.
Arm/Group | ASPIRE Group | GSA-ASPIRE-Network Group
All-Cause Mortality (participants affected / at risk) | 0/153 | 0/240
Serious Adverse Events (participants affected / at risk) | 0/153 | 0/240
Other Adverse Events (participants affected / at risk) | 0/153 | 0/240

LIMITATIONS AND CAVEATS:
This study faced some limitations including a low retention rate due to the timing of data collection, a lack of long-term behavioral data, and the reliance on staff for program delivery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-04): https://cdn.clinicaltrials.gov/large-docs/97/NCT02703597/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-24): https://cdn.clinicaltrials.gov/large-docs/97/NCT02703597/ICF_001.pdf